CLINICAL TRIAL: NCT06196840
Title: A Phase 2, Randomized Controlled, Open-Label Study to Establish the Safety and Efficacy of LX102 in Patients With Neovascular Age-related Macular Degeneration (nAMD) (VENUS)
Brief Title: Safety and Efficacy of LX102 Gene Therapy in Patients With Neovascular Age-related Macular Degeneration (nAMD) (VENUS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNOSTELLAR-LX102A01-2
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Neovascular Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; AMD; Neovascular AMD; Neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LX102 Dose 1 (Experimental): LX102 will be administered at the assigned dose level as a single dose subretinal injection on Day 0
  Interventions: Genetic: LX102 subretinal injection
- LX102 Dose 2 (Experimental): LX102 will be administered at the assigned dose level as a single dose subretinal injection on Day 0
  Interventions: Genetic: LX102 subretinal injection
- Control group (Active Comparator): Aflibercept at a fixed regimen will be administered.
  Interventions: Biological: Aflibercept intravitreal injection

INTERVENTIONS:
Genetic: LX102 subretinal injection — LX102: AAV-based gene therapy comprised of codon-optimized sequence encoding VEGF-trap
  Arms: LX102 Dose 1; LX102 Dose 2
Biological: Aflibercept intravitreal injection — Commercially available Active Comparator
  Arms: Control group

SUMMARY:
The goal of this study is to evaluate the overall safety and efficacy of LX102 gene therapy for nAMD.

DETAILED DESCRIPTION:
In this Phase 2, multi-center, randomized controlled study, subjects will be randomized to receive one of the two dose levels of LX102 (n=20 for each dose level), or aflibercept (n=10).

Safety, tolerability, and efficacy will be evaluated for a period of approximately 1 year from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent, and willing to attend follow-up visits.
2. Age ≥ 50, and ≤ 89.
3. Diagnosis of active CNV secondary to neovascular AMD.
4. BCVA ETDRS letters between 19 and 73.
5. Demonstrated a meaningful response to anti-VEGF therapy.

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to diseases other than nAMD.
2. Retinal detachment, uveitis, uncontrolled glaucoma in the study eye, or any condition preventing visual acuity improvement.
3. Absence of RPE tear at Screening.
4. Acute coronary syndrome, myocardial infarction or coronary artery revascularization, CVA, TIA in the last 6 months.
5. Uncontrolled hypertension defined as average SBP ≥160 mmHg or an average DBP ≥100 mmHg.
6. Uncontrolled diabetes defined as HbA1c >8.0%.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Best Corrected Visual Acuity (BCVA) | 36 weeks
  BCVA measured by ETDRS

SECONDARY OUTCOMES:
Mean change from baseline in Best Corrected Visual Acuity (BCVA) | 52 weeks
  BCVA measured by ETDRS
Mean change in Central Subfield Thickness (CST) from Baseline | 36 weeks, 52 weeks
  CST measured by spectral domain optical coherence tomography (SD-OCT)
Durability of LX102 treatment | 52 weeks
  Mean time from LX102 administration to anti-VEGF rescue injection for the first time, percentage of participants requiring anti-VEGF rescue injection, and mean number of anti-VEGF rescue injections through 52 weeks following LX102 administration.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 36 weeks, 52 weeks
  Incidence of ocular and systemic adverse events (AEs) and serious adverse events (SAEs) following LX102 subretinal injection

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Zhejiang University Eye Hospital, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Guangzhou Aier Eye Hospital, Guangzhou
  - Zhongshan Ophthalmic Center of Sun Yat-Sen University, Guangzhou
  - Shanghai Eye and ENT Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanxi Eye Hospital, Taiyuan
  - Tianjin Medical University Eye Hospital, Tianjin
  - Xuzhou No.1 People's Hospital, Xuzhou

IPD SHARING:
Plan to Share IPD: No